CLINICAL TRIAL: NCT06985589
Title: Efficacy and Safety of Fire Needle Therapy Combined With Cortex Phellodendri Compound Fluid Wet Compress for Acute Herpes Zoster: a Randomized Controlled Trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025514
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Acute Herpes Zoster
Keywords: acute Herpes zoster; fire needle therapy; Cortex Phellodendri compound fluid; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treated group (Experimental): The patients received fire needle (5 sessions, every other day) combined with CPCF wet compress treatment (3 times/day, 10 days) in addition to the basic treatment of the control group.
  Interventions: Procedure: Fire needle; Drug: Cortex Phellodendri compound fluid wet compress; Drug: basic treatment
- control group (Experimental): The control group received basic treatment, which consisted of penciclovir 0.5g/time per day intravenously, mecobalamin 0.5mg/time three times a day orally and pregabalin 75mg/time twice a day orally for 10 days.
  Interventions: Drug: basic treatment

INTERVENTIONS:
Procedure: Fire needle — At the beginning of the fire needle therapy, the patient was instructed to exposure the lesion in a comfortable position. And the Ashi point (lesion area) was disinfected with iodophor. The 95% alcohol lamp was lit and held by the left hand. Then the needle was held by the right hand in the outer flame of the alcohol lamp to heat the needle body, making the tip of the needle whiten. Subsequently, the needle was quickly and accurately puncted into the base of the herpes at a depth of about 2-5 mm, straight in and out. According to the number of herpes, the early-onset herpes was puncted first, and about 5 to 10 blisters were selected for each puncture. The acupuncture was performed 1-5 times according to the size of the herpes. The treatment was performed once every other day for total 5 sessions.
  Arms: treated group
Drug: Cortex Phellodendri compound fluid wet compress — For the Chinese herbal wet compress treatment, CPCF (Shandong Hanfang Pharmaceutical Co., LTD.) was decocted using forsythia, honeysuckle, phellodendron, dandelion, and centipede. Appropriate amount of liquid was diluted with 5 times the volume of water. Then according to the area of skin lesions, several pieces of medical fat-free cotton gauze with thickness of 8 layers were put into the liquid completely wet. After wringing out to a semi-dry state, the gauze was applied to the lesion for 15 minutes/time, 3 times a day, for 10 days.
  Arms: treated group
Drug: basic treatment — The basic treatment consisted of penciclovir 0.5g/time per day intravenously, mecobalamin 0.5mg/time three times a day orally and pregabalin 75mg/time twice a day orally for 10 days.

SUMMARY:
Herpes zoster (HZ) results from a reactivation of varicella-zoster virus (VZV), which causes primary infection leading to chickenpox and remains latent in the ganglia. Fire needle therapy is a non-pharmacological treatment that combines heat therapy with traditional acupuncture. This technique involves heating sterilized needles and swiftly inserting them into specific points or areas of the skin. Chinese herbal wet compress therapy is directly delivering medications to the lesion site, facilitating rapid transdermal absorption. This method ensures stable local drug concentrations and effectively alleviates pain, swelling, and other clinical symptoms. In this study, we conducted a randomized controlled trial to evaluate the clinical efficacy and safety of fire needle therapy combined with CPCF wet compress for the treatment of acute HZ. 32 acute HZ patients were randomized into control (standard antiviral and analgesic therapy) and treated groups (standard therapy plus fire needle [5 sessions, every other day] and CPCF wet compress [3 times/day, 10 days]). After 10 days of treatment, fire needle combined with CPCF wet compress significantly enhances symptom relief, pain reduction, and quality of life in acute HZ, with favorable safety.

DETAILED DESCRIPTION:
Herpes zoster (HZ) results from a reactivation of varicella-zoster virus (VZV), which causes primary infection leading to chickenpox and remains latent in the ganglia. Fire needle therapy is a non-pharmacological treatment that combines heat therapy with traditional acupuncture. This technique involves heating sterilized needles and swiftly inserting them into specific points or areas of the skin. Chinese herbal wet compress therapy is directly delivering medications to the lesion site, facilitating rapid transdermal absorption. This method ensures stable local drug concentrations and effectively alleviates pain, swelling, and other clinical symptoms. In this study, we conducted a randomized controlled trial to evaluate the clinical efficacy and safety of fire needle therapy combined with CPCF wet compress for the treatment of acute HZ. 32 acute HZ patients were randomized into control (standard antiviral and analgesic therapy) and treated groups (standard therapy plus fire needle [5 sessions, every other day] and CPCF wet compress [3 times/day, 10 days]). After 10 days of treatment, fire needle combined with CPCF wet compress significantly enhances symptom relief, pain reduction, and quality of life in acute HZ, with favorable safety.

ELIGIBILITY:
Inclusion Criteria:

1. males and females, aged 18-80 years old;
2. diagnosed as acute HZ with the course of disease within 7 days;
3. without history of other treatment before enrollment.

Exclusion Criteria:

1. specific types of HZ, including Ramsay Hunt Syndrom, ophthalmic, disseminated, deep, purpuric and central nervous system HZ;
2. pregnancy and lactation;
3. allergic to the related Chinese herbals;
4. patients with contraindications to penciclovir, mecobalamin and pregabalin; (e) history of hypertrophic scar or keloid;

(f) severe cardiovascular, cerebrovascular, digestive, urinary or hematopoietic disease; (g) mental disease; (h) coagulation disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
herpes zoster symptom and sign quantitative scoring scale | From enrollment to day 10
  The degree of the clinical symptoms and signs of HZ (including local pain, local itching, burning sensation, papular erythema, number of blisters, number of blister clusters, herpes character, ulcer, fever, local lymph node enlargement, and skin lesion area change) were divided into four grades: 0 (none), 1 (mild), 2 (moderate), and 3 (severe).
lesion improvement index n | From enrollment to day 10
  The lesion improvement index n was calculated by the formula: n (%) = (symptom and sign quantitative score at baseline - symptom and sign quantitative score at 10 days)/symptom and sign quantitative score at baselin ×100%.
the total improved rate | From enrollment to day 10
  The clinical improvement was graded as follows: clinical cure (n≥90%), significant improvement (70%≤n<90%), moderate improvement (30%≤n<70%), no improvement (n < 30%). The total improved rate was calculated as cases of (clinical cure + significant improvement + moderate improvement)/total cases×100%.

SECONDARY OUTCOMES:
questionnaire of Dermatology Life Quality Index | From enrollment to day 10
Pittsburgh sleep quality index | From enrollment to day 10
Hamilton Anxiety Scale | From enrollment to day 10
Visual analog scale | From enrollment to day 10
  The pain intensity due to HZ was evaluated by a visual analog scale (VAS) ranging from 0 to 10 (0: no pain, 1-3: mild, 4-6: moderate, 7-10: severe) at day 0 and day 10.
incidence of postherpetic neuralgia | From enrollment to day 90
  The incidence of postherpetic neuralgia was analysed at day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng JC, Liao YZ, Li JJ, Lu LH, Li HZ, Lu LM, Li QJ, Li LX, Wang SX, Lin GH. [Clinical efficacy of fire needling combined with cupping therapy on herpes zoster of acute stage and the effect on Th17/Treg cellular immune balance]. Zhongguo Zhen Jiu. 2023 Oct 12;43(10):1128-33. doi: 10.13703/j.0255-2930.20221005-k0004. Chinese. PMID 37802518
- [Background] Zhang Y, Li SH, Yang L, Xu QN, Pei WY, Liang ZH, Liu XH, Yang JJ, Lin GH. [Shallow Fire-needle Acupuncture Stimulation Plus Cupping Relieves Neuralgia and Down-regulates Serum Substance P Level in Patients with Acute Herpes Zoster]. Zhen Ci Yan Jiu. 2018 Aug 25;43(8):492-4. doi: 10.13702/j.1000-0607.170923. Chinese. PMID 30232851
- [Background] Huang SX, Mao M, Pu JJ, Chen YH, Deng L, Zhao H, Geng MJ, Zhong RF, Guo YJ, Liu ZS, Wang YH, Ye YM, Liu J, Yang T, Zhao AM, Chen XH, Zhu HY, Du YC. [Clinical research on fire filiform needle combined with mild moxibustion for postherpetic neuralgia]. Zhongguo Zhen Jiu. 2014 Mar;34(3):225-9. Chinese. PMID 24843959
- [Background] Chen J, Luo C, Ju P, Tu S, Shi S, Wang Z, Wu H. A bibliometric analysis and visualization of acupuncture and moxibustion therapy for herpes zoster and postherpetic neuralgia. Skin Res Technol. 2024 Jun;30(6):e13815. doi: 10.1111/srt.13815. PMID 38924142
- [Background] Dai YX, Yeh FY, Shen YJ, Tai YH, Huang N, Chang YT, Chen TJ, Li CP, Wu CY. Cigarette smoking and risk of herpes zoster: a population-based cohort study in Taiwan. Clin Exp Dermatol. 2021 Oct;46(7):1293-1298. doi: 10.1111/ced.14650. Epub 2021 May 11. PMID 33763912
- [Background] Patil A, Goldust M, Wollina U. Herpes zoster: A Review of Clinical Manifestations and Management. Viruses. 2022 Jan 19;14(2):192. doi: 10.3390/v14020192. PMID 35215786